CLINICAL TRIAL: NCT03900377
Title: A Multicenter, Open-label, Phase I/II Study to Investigate the Safety and Tolerability of SyB L-0501RI (Bendamustine Hydrochloride for Injection) Administered As an Intravenous (IV) Rapid Infusion Over 10 Minutes
Brief Title: Phase I/II Study of SyB L-0501RI in Combination With Rituximab to Treat Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018001
Record Dates: First submitted 2019-03-06; First posted 2019-04-03 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma, B-cell, Diffuse
Keywords: Lymphoma, B-cell, Diffuse, SyB L-0501RI
MeSH Terms: conditions — Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lg-B-NHL or MCL (Experimental): For previously untreated patients with Lg-B-NHL or MCL, rituximab will be intravenously administered at 375 mg/m^2 on Day 0 (the day before Day 1 only in Cycle 1), and SyB L-0501RI will be intravenously administered at 90 mg/m^2/day on Day 1 and Day 2 of each 28-day cycle with up to 6 cycles.
  Interventions: Drug: SyB L-0501RI
- DLBCL (Experimental): For patients with recurrent or refractory DLBCL, rituximab will be intravenously administered at 375 mg/m^2 on Day 1, and SyB L-0501RI will be intravenously administered at 120 mg/m^2/day on Day 2 and Day 3 of each 21-day cycle with up to 6 cycles.
  Interventions: Drug: SyB L-0501RI

INTERVENTIONS:
Drug: SyB L-0501RI — The specified dose of SyB L-0501RI and rituximab will be administered by intravenous rapid infusion over 10 minutes on specified days.
  Other Names: Rituximab

SUMMARY:
For SyB L-0501RI administered by an intravenous rapid infusion in combination with rituximab, the safety will be investigated in previously untreated patients with low-grade B-cell non-Hodgkin's lymphoma (Lg-B-NHL) or mantle cell lymphoma (MCL), and the safety and tolerability will be investigated in patients with recurrent/refractory diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
For previously untreated patients with Lg-B-NHL or MCL

Inclusion Criteria

Patients who satisfy all of the conditions listed below:

▪ Patients who satisfy all of the following criteria A) to D): A) Patients who are histopathologically confirmed to have one of the following subtypes of CD20 (cluster of differentiation 20)-positive Lg-B-NHL or MCL (excluding transformed lymphoma) by lymph node biopsy or evaluable tissue biopsy (World Health Organization [WHO] histological classification [4th edition]).

* Small lymphocytic lymphoma
* Splenic marginal zone lymphoma
* Lymphoplasmacytic lymphoma
* Extranodal marginal zone lymphoma of mucosa-associated lymphoid tissue (MALT)
* Nodal marginal zone lymphoma
* Follicular lymphoma (Grade 1, 2, 3a)
* MCL B) Patients who have at least one measurable lesion (>1.5 cm in major axis on computed tomography [CT]).

C) Patients without a history of treatment for lymphoma. D) Patients with at least one of the following clinical signs or symptoms (with the exception of MCL patients).

1. Bulky disease >7 cm in major axis on CT (excluding lesions in the spleen)
2. B symptoms

   * Unexplained fever exceeding 38.0ºC
   * Night sweats
   * Weight loss of more than 10% within 6 months before registration
3. Elevated serum lactate dehydrogenase (LDH) or β2-microglobulin level
4. Involvement of at least 3 regional lymph nodes >3 cm in major axis on CT
5. Symptomatic splenomegaly
6. Compressive symptoms
7. Pleural effusion and/or ascites

   * Patients aged between 20 and 79 years (at the time of registration).
   * Patients who are expected to survive for at least 3 months.
   * Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2.
   * Patients with adequate functional reserve of major organs (bone marrow, heart, lungs, liver, kidneys, etc.).

     * Neutrophil count: ≥1,500/mm^3
     * Platelet count: ≥75,000/mm^3
     * Aspartate aminotransferase (AST) [glutamic oxaloacetic transaminase [GOT]): ≤3.0 times the institution's upper limit of normal (ULN)
     * Alanine aminotransferase (ALT) [glutamic pyruvic transaminase (GPT)]: ≤3.0 times the institution's ULN
     * Total bilirubin: <2.0 mg/dL
     * Serum creatinine: <2.0 mg/dL
     * Percutaneous arterial oxygen saturation (SpO2): ≥95% or Partial arterial oxygen pressure (PaO2): ≥65 mmHg
     * No abnormal findings requiring treatment on electrocardiogram (ECG)
     * Left ventricular ejection fraction (LVEF) on echocardiography: ≥55%
   * Patients who have provided written informed consent to participate in this study.

Exclusion Criteria

Patients who meet any of the following conditions will be excluded:

* MCL patients aged ≤65 years (at the time of registration).
* Patients who have a history of treatment for Lg-B-NHL or MCL (chemotherapy, radiotherapy, antibody therapy or antitumor steroid therapy).
* Patients who have previously received hematopoietic stem cell transplantation.
* Patients with invasion to central nervous system (CNS) or clinical symptoms suspected of CNS invasion.
* Patients with serious active infection (requiring antibiotic, antifungal, or antiviral IV injection).
* Patients with serious complications (such as hepatic failure and renal failure).
* Patients with concurrent or previous, serious cardiac disease (e.g., myocardial infarction, ischemic heart disease); however, patients with arrhythmias are allowed to be enrolled if it does not require treatment at the time of registration.
* Patients with serious gastrointestinal symptoms (such as high-grade or severe nausea/vomiting or diarrhea).
* Patients with malignant pleural effusion, pericardial effusion, or ascites.
* Patients positive for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody (patients with positive hepatitis B virus [HBV]-DNA quantitative test results if they are negative for HBs antigen and positive for HBs antibody or hepatitis B core [HBc] antibody).
* Patients with serious bleeding tendencies (such as disseminated intravascular coagulation [DIC]).
* Patients with a fever of 38.0ºC or higher (with the exception of fever developing as a B symptom).
* Patients with concurrent or previous interstitial pneumonia, pulmonary fibrosis, or chronic obstructive pulmonary disease.
* Patients with active multiple primary cancers or patients with a history of other malignancy within the past 5 years, with the exception of basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or digestive organs.
* Patients with concurrent or previous autoimmune hemolytic anemia.
* Patients who have previously received bendamustine hydrochloride.
* Patients who have received a cytokine preparation, such as granulocyte colony- stimulating factor (G-CSF) or erythropoietin, or blood transfusions within 2 weeks before a screening test for this study.
* Patients who have received other investigational products or unapproved drugs within 3 months before registration for this study.
* Patients with a history of allergy to medications similar to SyB L-0501RI (e.g., alkylating agents and purine-nucleoside derivatives).
* Patients who cannot tolerate rituximab.
* Pregnant, possibly pregnant, or lactating women.
* Patients, whether male or female, who do not agree to use contraception.

Duration:

Male patients; during the treatment period and for 6 months after treatment Female patients with no menstruation; during the treatment period Female patients with menstruation; during the treatment period and for 3 months after treatment

* Patients with drug addiction, narcotic addiction, or alcohol dependence.
* Patients who are unable to take pre-treatment medication due to drug allergies or the like.
* Patients who are otherwise judged by the investigator or subinvestigator to be unsuitable as a subject.

For patients with recurrent or refractory DLBCL

Inclusion Criteria

Patients who satisfy all of the conditions listed below:

▪ Patients who satisfy both of the following criteria A and B: A) Patients who are histopathologically confirmed to have CD20-positive DLBCL (excluding transformed lymphoma) by lymph node biopsy or evaluable tissue biopsy (WHO histological classification [4th edition]).

B) Patients with recurrent or refractory DLBCL who have had disease progression after standard rituximab plus cyclophosphamide, doxorubicin, vincristine and prednisolone (R-CHOP) therapy or R-CHOP-like therapy as first-line treatment.

* Patients aged between 20 and 79 years (at the time of registration).
* Patients who are expected to survive for at least 3 months.
* Patients with an ECOG PS of 0 to 2.
* Patients with adequate functional reserve of major organs (bone marrow, heart, lungs, liver, kidneys, etc.).

  * Neutrophil count: ≥1,500/mm^3
  * Platelet count: ≥75,000/mm^3
  * AST (GOT): ≤3.0 times the institution's ULN
  * ALT (GPT): ≤3.0 times the institution's ULN
  * Total bilirubin: <2.0 mg/dL
  * Serum creatinine: <2.0 mg/dL
  * SpO2: ≥95% or PaO2: ≥65 mmHg
  * No abnormal findings requiring treatment on ECG
  * LVEF on echocardiography: ≥55%
* Patients who have provided written informed consent to participate in this study.

Exclusion Criteria

Patients who meet any of the following conditions will be excluded:

* Patients with an off-treatment interval of less than 3 weeks between the last day of preceding treatment (chemotherapy, radiotherapy, antibody therapy, or antitumor steroid therapy) for DLBCL and the day of registration for this study.
* Patients who are judged by the investigator or subinvestigator to be suitable for autologous peripheral blood stem cell transplantation.
* Patients who have previously received allogeneic hematopoietic stem cell transplantation.
* Patients who have previously received radioimmunotherapy
* Patients with invasion to CNS or clinical symptoms suspected of CNS invasion.
* Patients with serious active infection (requiring antibiotic, antifungal, or antiviral IV injection).
* Patients with serious complications (such as hepatic failure and renal failure).
* Patients with concurrent or previous, serious cardiac disease (e.g., myocardial infarction, ischemic heart disease); however, patients with arrhythmias are allowed to be enrolled if it does not require treatment at the time of registration.
* Patients with serious gastrointestinal symptoms (such as high-grade or severe nausea/vomiting or diarrhea).
* Patients with malignant pleural effusion, pericardial effusion, or ascites.
* Patients positive for HBs antigen, HCV antibody, or HIV antibody (patients with positive HBV-DNA quantitative test results if they are negative for HBs antigen and positive for HBs antibody or HBc antibody).
* Patients with serious bleeding tendencies (such as DIC).
* Patients with a fever of 38.0ºC or higher (with the exception of fever developing as a B symptom).
* Patients with concurrent or previous interstitial pneumonia, pulmonary fibrosis, or chronic obstructive pulmonary disease.
* Patients with active multiple primary cancers or patients with a history of other malignancy within the past 5 years, with the exception of basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or digestive organs.
* Patients with concurrent or previous autoimmune hemolytic anemia.
* Patients who have previously received bendamustine hydrochloride.
* Patients who have received a cytokine preparation, such as G-CSF or erythropoietin, or blood transfusions within 2 weeks before a screening test for this study.
* Patients who have received other investigational products or unapproved drugs within 3 months before registration for this study.
* Patients with a history of allergy to medications similar to SyB L-0501RI (e.g., alkylating agents and purine-nucleoside derivatives).
* Patients who cannot tolerate rituximab.
* Pregnant, possibly pregnant, or lactating women.
* Patients, whether male or female, who do not agree to use contraception.

Duration:

Male patients; during the treatment period and for 6 months after treatment Female patients with no menstruation; during the treatment period Female patients with menstruation; during the treatment period and for 3 months after treatment

* Patients with drug addiction, narcotic addiction, or alcohol dependence.
* Patients who are unable to take pre-treatment medication due to drug allergies or the like.
* Patients who are otherwise judged by the investigator or subinvestigator to be unsuitable as a subject.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Adverse events (type, frequency, severity) | Up to 36 weeks
Number of subjects with adverse event | Up to 36 weeks
Number of adverse events | Up to 36 weeks
Number of subjects with abnormality (Common Terminology Criteria for Adverse Events [CTCAE] grade ≥3) in laboratory test values | Up to 36 weeks
Number of subjects with grade ≥3 physical examination finding | Up to 36 weeks
Number of subjects with dose limiting toxicity in DLBCL arm | Up to 36 weeks

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 36 weeks
Overall response rate (antitumor effect : ≥ partial response [PR]) | Up to 36 weeks
Progression-free survival (PFS) | Up to 36 weeks
The maximum concentration (Cmax) of unchanged SyB L-0501 | Prior to and 5, 10 min after start of administration, and 5, 15, 30, 60, 120, 240, 360 min after completion of administration on Day 1 of the 1st cycle in Lg-B-NHL or MCL Arm (in DLBCL Arm, Day 2 of the 1st cycle)
The maximum drug concentration time (Tmax) of unchanged SyB L-0501 | Prior to and 5, 10 min after start of administration, and 5, 15, 30, 60, 120, 240, 360 min after completion of administration on Day 1 of the 1st cycle in Lg-B-NHL or MCL Arm (in DLBCL Arm, Day 2 of the 1st cycle)
The area under the curve (AUC) for unchanged SyB L-0501 | Prior to and 5, 10 min after start of administration, and 5, 15, 30, 60, 120, 240, 360 min after completion of administration on Day 1 of the 1st cycle in Lg-B-NHL or MCL Arm (in DLBCL Arm, Day 2 of the 1st cycle)
The half-life period (T1/2) of unchanged SyB L-0501 | Prior to and 5, 10 min after start of administration, and 5, 15, 30, 60, 120, 240, 360 min after completion of administration on Day 1 of the 1st cycle in Lg-B-NHL or MCL Arm (in DLBCL Arm, Day 2 of the 1st cycle)

CONTACTS AND LOCATIONS:
Locations (14):
- Japan (14):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Ōta, Gunma
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Isehara, Kanagawa
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Koto-ku, Tokyo
  - Research Site, Akita
  - Research Site, Fukuoka
  - Research Site, Kagoshima
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Okayama
  - Research Site, Yamagata

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ishizawa K, Yokoyama M, Kato H, Yamamoto K, Makita M, Ando K, Ueda Y, Tachikawa Y, Suehiro Y, Kurosawa M, Kameoka Y, Nagai H, Uoshima N, Ishikawa T, Hidaka M, Ito Y, Utsunomiya A, Fukushima K, Ogura M. A phase I/II study of 10-min dosing of bendamustine hydrochloride (rapid infusion formulation) in patients with previously untreated indolent B-cell non-Hodgkin lymphoma, mantle cell lymphoma, or relapsed/refractory diffuse large B-cell lymphoma in Japan. Cancer Chemother Pharmacol. 2022 Jul;90(1):83-95. doi: 10.1007/s00280-022-04442-2. Epub 2022 Jul 7. PMID 35796785